CLINICAL TRIAL: NCT05604599
Title: Intranasal Premedication With Dexmedetomidine Versus Intravenous Dexmedetomidine for Hypotensive Anesthesia During Functional Endoscopic Sinus Surgery in Adults: A Randomized Triple-Blind Trial
Brief Title: Intranasal Versus Intravenous Dexmedetomidine for Hypotensive Anesthesia in FESS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Neveen Abd El Maksoad Kohaf, Lecturer of Clinical Pharmacy, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB 00012367-22-011-001
Record Dates: First submitted 2022-10-28; First posted 2022-11-03 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Functional Endoscopic Sinus Surgery; Premedication; Analgesia
Keywords: Dexmedetomidine; Intranasal; Intravenous
MeSH Terms: conditions — Agnosia | interventions — Propofol; Fentanyl; Isoflurane; Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal dexmedetomidine group (Active Comparator): 30 patients will receive 1µg/kg dexmedetomidine diluted in 10ml 0.9% saline intranasally preoperative administered to each naris as drops 45 -60 min before the operation +infusion saline.
  Interventions: Drug: Intranasal dexmedetomidine
- Intravenous dexmedetomidine group (Active Comparator): 30 patients will receive a dose of dexmedetomidine 1 µg/kg diluted in 10ml 0.9% saline infused over 45- 60 min before induction of anesthesia + intranasal saline.
  Interventions: Drug: Intravenous dexmedetomidine

INTERVENTIONS:
Drug: Intranasal dexmedetomidine — 45 -60 min before the operation, patients will receive dose of dexmedetomidine 1microgram/kg diluted in 10ml 0.9% saline administered to each naris as drops + infusion saline
  Other Names: Propofol 2 mg/kg; fentanyl 1 µg/kg; Cis-atracurium 0.15mg / kg; Isoflurane 1-1.5% in 50% oxygen
  Arms: Intranasal dexmedetomidine group
Drug: Intravenous dexmedetomidine — patients will receive loading dose of dexmedetomidine 1 µg/kg diluted in 10ml 0.9% saline infused over 45- 60 min before induction of anesthesia, followed by continuous infusion of (0.4 µ g/kg/h) + intranasal saline.
  Other Names: Propofol 2 mg/kg,, fentanyl 1 µg/kg , Cis-atracurium 0.15mg / kg and Isoflurane 1-1.5% in 50% oxygen
  Arms: Intravenous dexmedetomidine group

SUMMARY:
Intranasal dexmedetomidine provided good pharmacokinetic profile. However, intravenous dexmedetomidine have been used in functional endoscopic sinus surgery for several outcomes, there is lack in studies that had compared the efficacy of intravenous and Intranasal Dexmedetomidine for improving quality of the operative field in functional endoscopic sinus surgery.

Therefore, we established this randomized study to compare intranasal dexmedetomidine with intravenous dexmedetomidine improving quality of the operative field in functional endoscopic sinus surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 21 years of age.
* Both genders.
* American Society of Anesthesiologists (ASA) physical status classification I - III who underwent functional endoscopic sinus surgery.

Exclusion Criteria:

* Patients with a body mass index > 30 kg/m2
* Existing or recent significant disease.
* Contraindications to the use of dexmedetomidine.
* History or presence of a significant disease.
* Significant cardiovascular disease risk factors.
* Significant coronary artery disease.
* Any known genetic predisposition.
* History of any kind of drug allergy.
* Drug abuse.
* Psychological or other emotional problems.
* Special diet or lifestyle.
* Clinically significant abnormal findings in physical examination, electrocardiographic (ECG) or laboratory screening.
* Known systemic disease requiring the use of anticoagulants.
* Any nasal disorders that may hinder nasal administration of the drugs as repeated nasal bleeding or nasal tumors.
* Patients with a history of previous functional endoscopic sinus surgery.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-03-05 (Actual); Study Completion 2023-03-05 (Actual)

PRIMARY OUTCOMES:
Improving quality of the operative field. | during surgery (intraoperatively) 2 hours
  Quality of intraoperative surgical field during functional endoscopic sinus surgery will be evaluated by the surgeons by rating the amount of bleeding according to a 6-point scale by Formmer's scores of surgical field quality (0= no bleeding; 1= bleeding, so mild it was not even a surgical nuisance; 2= moderate bleeding, a nuisance but without interference; 3= moderate bleeding that moderately compromised surgical; 4= bleeding, heavy but controllable, that significantly interfered; 5= massive uncontrollable bleeding.
Amount of atropine consumption | First 24 hours postoperatively
  The total amount of atropine consumed will be recorded

SECONDARY OUTCOMES:
Hemodynamics(Heart rate (bpm)) | 2 hours
  Heart rate (bpm), at base line, 5minute, 10 minute , 30 minute, 45 minute, 60 minute after patient received intranasal and after infusion of loading dose of dexmedetomidine , 5, 15, 30, 45, 60 minutes after induction of anesthesia, at end of surgery and 30 minute after recovery.
Hemodynamics(Mean arterial blood pressure mm Hg)) | 2 hours
  Mean arterial blood pressure mm Hg) at base line, 5minute, 10 minute , 30 minute, 45 minute, 60 minute after patient received intranasal and after infusion of loading dose of dexmedetomidine , 5, 15, 30, 45, 60 minutes after induction of anesthesia, at end of surgery and 30 minute after recovery.
Pain score | First 24 hours postoperatively
  Pain measured with VAS: (visual analogue scale) will be assessed in post anesthesia care unit, 1, 2, 4, 6, 8, 12, 18, and 24hours postoperative.
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). patients are asked to rate their current level of pain by placing a mark on the line.
Adverse events | 24 postoperatively
  Adverse events will be recorded such as nausea, vomiting, hypotension and bradycardia.
hemostatic stuffing | 24 hours postoperatively
  The degree of adverse reactions of hemostatic stuffing after functional endoscopic sinus surgery will be also evaluated (1=no swelling, can tolerate; 2= swelling, can barely tolerate; 3= swelling, cannot tolerate).

CONTACTS AND LOCATIONS:
Locations (1):
- Facualty of Medicine(Damietta), Al Azhar University, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
data can be shared with a reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP